CLINICAL TRIAL: NCT04940806
Title: The Value of Combined Detection of Orexin-A, HLA Gene, PSG and MSLT in the Evaluation of Patients With Narcolepsy
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Qianfoshan Hospital (Other)
Responsible Party: Principal Investigator, Lili Cao, Professor, Qianfoshan Hospital
Other Study IDs: QianfoshanH H
Record Dates: First submitted 2021-06-15; First posted 2021-06-28 (Actual); Last update posted 2021-06-28 (Actual); Status verified 2021-06

CONDITIONS: Narcolepsy
Keywords: Narcolepsy; Orexin; HLA gene; Polysomnography; Multiple sleep latency test
MeSH Terms: conditions — Narcolepsy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 120 patients with narcolepsy

SUMMARY:
By comparing the differences of orexin-A, HLA gene, PSG, MSLT and other parameters in the evaluation of narcolepsy patients, investigators could find out the relatively high value indicators in the diagnosis of narcolepsy, which is helpful to guide the clinical discovery, diagnosis and treatment of narcolepsy.

DETAILED DESCRIPTION:
Narcolepsy is a lifelong sleep disorder disease, mainly occurs in the 15~30 year old youth. The incidence rate in different country population is different, which is 0.04% in China. Because of its low incidence rate, and the lack of clinicians' knowledge, it is easy to cause missed diagnosis and misdiagnosis. The decrease of cerebrospinal fluid orexin-A level, positive HLA-DQB1 * 0602 and MSLT all have directive significance for the diagnosis of narcolepsy, but patients with other diseases and healthy people can also show positive indicators. These false positives may lead to wrong judgments. By comparing the differences of orexin-A, HLA gene, PSG, MSLT and other parameters in the evaluation of narcolepsy patients, investigators could find out the relatively high value indicators in the diagnosis of narcolepsy, which is helpful to guide the clinical discovery, diagnosis and treatment of narcolepsy.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 10-70 years old;
2. The symptoms lasted for at least 3 months;
3. With or without cataclysm;
4. MSLT showed that the sleep latency was less than or equal to 8 min, there were two or more times of sleep, the onset of REM sleep;
5. Somnolence can not be explained by other diseases, such as insufficient sleep, OSAHS, delayed sleep phase, drug or drug use, etc.

Exclusion Criteria:

1. Somnolence was caused by sleep disorders, central nervous system diseases, brain trauma and other non narcolepsy;
2. Recent lack of sleep or irregular sleep;
3. PSG and MSLT examination can not be diagnosed as narcolepsy;
4. Poor compliance, taking drugs or food and beverage containing central inhibitory components during the trial;
5. Severe neuropsychiatric disorders can not cooperate with the examination;
6. Patients with history of rheumatism, diabetes, ankylosing spondylitis and other HLA related diseases.

Ages: 10 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The participants of the study were patients who were admitted to the sleep center of Qianfoshan Hospital of Shandong Province from August 2019 to June 2025. All patients had clinical symptoms of narcolepsy and were diagnosed as narcolepsy by auxiliary laboratory examination.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2021-05-01 (Actual); Primary Completion 2024-05 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Pittsburgh sleep quality index scale | 1 day
  The sleep quality of the patients in the past month was evaluated. The higher the score, the worse the sleep quality. The scale of the score is 0-21, and the higher score means a worse outcome.
Epworth Sleeping Scale | 1 day
  Assess the possibility of dozing (not just feeling tired) in recent months. The higher the score was, the more likely it was to doze during the day. The scale of the score is 0-24, and the higher score means a worse outcome.
Insomnia Severity Index | 1 day
  Liker scale is used to evaluate the nature and symptoms of sleep disorders. The higher the score, the more serious the insomnia. The scale of the score is 0-28, and the higher score means a worse outcome.
Ullanlinna Narcolepsy Scale | 1 day
  It can be effectively distributed as a control group for sleeping sickness and healthy people. The total score is between 0-44. The higher the score is, the higher the possibility of narcolepsy is. The scale of the score is 0-44, and the higher score means a worse outcome.
Stanford Sleepiness Scale | 1 day
  Subjective assessment tool to assess sleepiness. The scale of the score is 0-7, and the higher score means a worse outcome.
Hamilton Anxiety Scale | 1 day
  It can be used to evaluate the depressive symptoms of depression, manic depression, neurosis and other diseases. The higher the score, the more anxiety.
  It can be used to evaluate the depressive symptoms of depression, manic depression, neurosis and other diseases. The higher the score, the more anxiety.
  It can be used to evaluate the depressive symptoms of depression, manic depression, neurosis and other diseases. The higher the score, the more anxiety.
  It can be used to evaluate the depressive symptoms of depression, manic depression, neurosis and other diseases. The higher the score, the more anxiety.
  It can be used to evaluate the depressive symptoms of depression, manic depression, neurosis and other diseases. The higher the score, the more anxiety.
  The scale of the score is 0-56, and the higher score means a worse outcome.
Hamilton Depression Scale | 1 day
  It can be used to evaluate the depressive symptoms of depression, manic depression, neurosis and other diseases. The higher the score, the more severe the depression. The scale of the score is 0-96, and the higher score means a worse outcome.
Montreal Cognitive Assessment Scale | 1 day
  A full score of 30 points, and ≥ 26 points were considered as normal cognition.
Polysomnography | 2 days
  The participants completed PSG in the sleep room from 10:00 p.m. to 6:00 a.m. the next day. The test lasted for at least 7 hours to ensure that the participants had enough sleep before MSLT. Professional and technical personnel interpreted the results and calculated the PSG sleep latency, REM latency, soremps sleep, sleep efficiency, AHI and the proportion of each sleep period.
Multiple sleep latency test | 1 day
  Participants completed MSLT in the sleep room, according to the standard method published by the American Sleep Society, 20 minutes each time, a total of 5 times.Professional and technical personnel interpreted the results and calculated the MSLT MSL, soremps sleep; In MSLT, MSL ≤ 8 min and soremps ≥ 2 were positive.
The level of orexin-A | 1 week
  The qualified clinician performed lumbar puncture on the participants, extracted cerebrospinal fluid and sub packed it into EP tube. The samples that could not be detected immediately were stored at - 80 ℃ for detection (about half a year for detection). The level of orexin-A in cerebrospinal fluid was detected by enzyme-linked immunosorbent assay (ELISA). CSF orexin-A concentration is either ≤ 110 pg/mL or <1/3 of mean values obtained in normal human with the same standardized assay.
Human leukocyte antigen gene | 1 week
  After blood sampling, HLA gene was detected by sequence specific primer gene amplification. Most ofl patients with cataplexy are positive for DQB1*0602, which is a HLA subtype.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Shandong First Medical University, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No